CLINICAL TRIAL: NCT03003650
Title: ACURATE TF™ Transfemoral Aortic Bioprosthesis for Implantation in Patients With Severe Aortic Stenosis:CE-approval Cohort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Symetis SA (Industry)
Responsible Party: Sponsor
Organization: Boston Scientific Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TF89
Record Dates: First submitted 2016-12-02; First posted 2016-12-28 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Symptomatic Aortic Stenosis
Keywords: Severe Symptomatic Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Symetis ACURATE TF™ (Experimental): Patient implanted with ACURATE TF™Bioprosthesis.
  Interventions: Device: ACURATE TF™

INTERVENTIONS:
Device: ACURATE TF™ — ACURATE TF™Transfemoral Aortic Bioprosthesis is intended for subjects with severe symptomatic Aortic Stenosis and are considered high risk for surgical conventional Aortic Valve Replacement .
  Other Names: ACURATE TF™Transfemoral Aortic Bioprosthesis and Delivery System

SUMMARY:
First clinical experience on the ACURATE TF™ Transfemoral Aortic Bioprosthesis Implantation in Patients with Severe Aortic Stenosis to collect human data pertaining to the safety and performance of the device from three different cohorts

DETAILED DESCRIPTION:
A prospective, multicenter, "CE-approval cohort" analysis with the Symetis ACURATE TF™ Transfemoral Aortic Bioprosthesis for minimal invasive implantation via transfemoral access to treat patients with severe aortic stenosis where conventional aortic valve replacement (AVR) via open heart surgery is considered to be associated with high risk, to evaluate the feasibility and performance of the implantation at 30-Days and at 1-Year Follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 75 years of age and older
2. Logistic EuroSCORE ≥ 20%
3. Severe aortic stenosis characterized by mean aortic gradient > 40 mmHg or peak jet velocity > 4.0 m/s or aortic valve area of < 1.0 cm2
4. New York Heart Association (NYHA) Functional Class > II
5. Aortic annulus diameter from ≥ 21mm up to ≤ 27mm by Trans-esophageal Echocardiography (TEE)
6. Patient not a surgical candidate due to significant co-morbid conditions unrelated to aortic stenosis
7. Patient willing to participate in the study and provide signed informed consent

Exclusion Criteria:

1. Unicuspid or bicuspid aortic valve
2. Extreme eccentricity of calcification
3. Severe mitral regurgitation ( >2+)
4. Pre-existing prosthetic heart valve in any position and / or prosthetic ring
5. Aortic or peripheral anatomy NOT appropriate for transfemoral implant
6. Thoracic (TAA) or abdominal (AAA) aortic aneurysm
7. Presence of endovascular stent graft for treatment of TAA or AAA
8. TEE is contraindicated
9. Left Ventricular Ejection Fraction (LVEF) < 30% by echocardiography (ECHO)
10. ECHO evidence of intracardiac mass, thrombus, or vegetation
11. Acute Myocardial Infarction (AMI) within 1 month prior to implant procedure
12. Percutaneous Coronary Intervention (PCI), except for balloon valvuloplasty (BAV) within 1 month prior to implant procedure
13. Previous Transien Ischemic Attack (TIA) or stroke within 3 months prior to implant procedure
14. Active ulcer or gastrointestinal (GI) bleeding within 3 months prior to implant procedure
15. Any scheduled surgical or percutaneous procedure to be performed prior to 30 day visit
16. History of bleeding diathesis or coagulopathy or refusal of blood transfusions
17. Systolic pressure <80 mmHg, cardiogenic shock, need for inotropic support or Intra-Aortic Balloon Pump (IABP)
18. Primary hypertrophic obstructive cardiomyopathy (HOCM)
19. Active infection, endocarditis or pyrexia
20. Hepatic failure
21. Chronic renal dysfunction with serum creatinine > 2.5 mg/dL or renal dialysis
22. Refusal of surgery
23. Severe Chronic Obstructive Pulmonary Disease (COPD) requiring home oxygen
24. Neurological disease severely affecting ambulation or daily functioning, or dementia
25. Life expectancy < 12 months due to non-cardiac co-morbid conditions
26. Known hypersensitivity/contraindication to study medication, contrast media, or nitinol
27. Currently participating in an investigational drug or another device study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 89 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Freedom from all-cause mortality | 30-Day Follow-up
  Rate of all-cause mortality

SECONDARY OUTCOMES:
Rate of MACCE (major cardiac and cerebrovascular event) related to the ACURATE TF™ Transfemoral Aortic Bioprosthesis and Delivery System. | 30-Days and 12 Months Follow-up
  Rate of major cardiac and cerebrovascular event (MACCE) at 30 days and at 12 months follow-up related to ACURATE TF™ Transfemoral Aortic Bioprosthesis and Delivery System and defined as all cause death, myocardial infarction, re-intervention and stroke.
Change in NYHA class over time | 30-Day and 12-Month
  Functional improvement from baseline NYHA classification at 30 day and at 12 month follow-up.
Procedural success during device implantation | intraoperative
  Procedural Success defined as stable study device placement at intended site and adequate device functioning immediately post-implantation, confirmed by angiography and echocardiography and without intra-procedural mortality.
Device success | 30-Day and 12-Month Follow-up
  Device success is defined as adequate functioning of the study device as confirmed by angiography and/or echocardiography.
  The following data points will be analyzed for adequate functioning of the study device:
  * Effective orifice area and index (EOA)
  * Peak jet velocity
  * Transvalvular aortic gradient (mean)
  * Paravalvular and intravalvular (central) leak
  * Aortic Insufficiency
  * Valve function and morphology

CONTACTS AND LOCATIONS:
Locations (6):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil
- Germany (4):
  - Kerckhoff Klinik GmbH, Bad Nauheim
  - Universitätsklinikum Bonn, Bonn
  - Herzzentrum Universitätsklinikum Köln, Cologne
  - Universitäres Herzzentrum Hamburg, Hamburg
- Osaka University Hospital, Osaka, Japan